CLINICAL TRIAL: NCT06058117
Title: PEGASUS: Paediatric European Group A Streptococcal United Study.
Brief Title: Paediatric European Group A Streptococcal United Study.
Acronym: PEGASUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Noordwest Ziekenhuisgroep (Other)
Collaborators: European Society for Paediatric Infectious Diseases (Other); Medical University of Graz (Other); University Hospital Munich (Other); National and Kapodistrian University of Athens (Other); Mitera Hospital (Other); Children's hospital Iceland (Unknown); University of Padova (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Riga Stradins University (Other); Maasstad Hospital (Other); HagaZiekenhuis (Other); Leiden University Medical Center (Other); Wroclaw Medical University (Other); University Medical Centre Ljubljana (Other); Hospital Clínico Universitario de Santiago de Compostela (Unknown); Hospital Universitario 12 de Octubre (Other); Hospital Universitario La Paz (Other); Gregorio Marañón Hospital (Other); Karolinska Institutet (Other); Imperial College London (Other); University of Liverpool (Other); Newcastle University (Other)
Responsible Party: Principal Investigator, Dorine Borensztajn, Principal investigator, MD, PhD, MSc., Noordwest Ziekenhuisgroep
Other Study IDs: 1.2
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Invasive Group A Beta-Haemolytic Streptococcal Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with invasive group A streptococcal disease: children with invasive group A streptococcal disease or other invasive or emergent infectious disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention, this is an observational study

SUMMARY:
Introduction Since 2022 there are reports of a rapid increase in invasive group A streptococcal infections (iGAS) in children in some but not all European countries. Detailed information on this increase is lacking. Furthermore, an increase in other invasive infections as well as the emergence of novel pathogens and disease entities is seen, such as MIS-C and severe hepatitis of unknown origin.

Aims To set up a European research network and describe the incidence, risk factors, clinical phenotypes, microbiology and resistance, treatment, and outcomes of iGAS in children across Europe. The network will subsequently be utilized for early alerting regarding the rise of other invasive and emerging infections in children. It will enable swift data collection pertaining to patient characteristics, presentation, progression, and treatment.

Methods International, retrospective cohort and observational surveillance study of children 0-18y attending the ED or admitted to the hospital with iGAS. Clinical and microbiological data, national vaccination schedules, and COVID non-pharmaceutical interventions (NPIs) will be collected and compared between countries. Subsequently, the network will be employed to raise alarms regarding the surge of other invasive infections or emerging infections in children. Anonymous data about these novel infections will be collected, similar to the data from iGAS (clinical characteristics and microbiological data). The study is a non-profit study.

Significance Our study will describe variation in the clinical phenotypes of iGAS, will aid in the understanding of its association with COVID NPIs and allow for comparison between countries. Furthermore, it will aid in early recognition of invasive and emergent infectious diseases in children and the reduction of outbreaks.

ELIGIBILITY:
* All children (1 month-18 years)
* attending the Emergency Department and/or admitted to the participating hospital - with iGAS infection or other invasive or emergent infectious disease.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Definitions
  Confirmed iGAS infection:
  * Clinical presentation consistent with iGAS* AND
  * Isolation of group A streptococcus by culture or PCR or antigen detection test from a normally sterile body site
  Probable iGAS infection:
  * Clinical presentation consistent with STSS or necrotizing fasciitis * AND
  * Isolation of group A streptococcus by culture or PCR or antigen detection test from a non-sterile body site AND
  * No evidence of other pathogen explaining the clinical presentation
    * Clinical presentation consistent with iGAS:
  Clinically severe illness, such as sepsis, septic shock, STSS, pneumonia, meningitis, arthritis, osteomyelitis, myositis or necrotizing fasciitis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
What is the incidence of iGAS in children before, during and after COVID NPIs in different European countries? | 2018-2025
Is there a change in clinical phenotypes and outcome during these periods? | 2018-2025

SECONDARY OUTCOMES:
Is there a change in emm types and other virulence factors during these periods | 2018-2025
Are there differences in antimicrobial resistance between periods and between 4. Are there differences in antimicrobial resistance between periods and between countries | 2018-2025
Can we identify risk factors for iGAS infection (e.g., preceding infections, age)? | 2018-2025
Can we explain differences between countries (e.g., differences in vaccination strategies, NPIs or emm types) | 2018-2025
Can we use this research network for early alarming on other invasive and emergent infectious diseases in children | 2018-2025

CONTACTS AND LOCATIONS:
Locations (1):
- Noordwest Ziekenhuisgroep, Alkmaar, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided